CLINICAL TRIAL: NCT03760211
Title: A Multisite Randomized Trial of Battle Viro: A Mobile Gaming App to Improve ART Adherence for Youth
Brief Title: A Mobile Gaming App to Improve ART Adherence for Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: University of Mississippi Medical Center (Other); Boston Medical Center (Other); Emory University (Other)
Responsible Party: Principal Investigator, Laura Whiteley, Assistant Professor, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 217318
Record Dates: First submitted 2018-11-19; First posted 2018-11-30 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2024-04

CONDITIONS: Medication Adherence; HIV/AIDS
MeSH Terms: conditions — Medication Adherence; Acquired Immunodeficiency Syndrome | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multilevel Gaming Adherence (Experimental): Participants in the intervention arm will receive Multilevel Gaming Adherence Intervention. Participants receive Battle Viro on their mobile phones, an electronic pill monitoring device, and, for 24 weeks, game-related text messages guided by medication adherence data (collected from an electronic pill monitoring device).
  Interventions: Behavioral: Multilevel Gaming Adherence Intervention
- Treatment as Usual + (Active Comparator): TAU+ participants will receive the Treatment As Usual + intervention, which includes receiving a non-HIV related mobile game and an electronic pill monitoring device.
  Interventions: Behavioral: Treatment as Usual +

INTERVENTIONS:
Behavioral: Multilevel Gaming Adherence Intervention — Combination of electronic medication monitoring device with Information-Motivation-Behavior based mobile gaming application tailored for those living with HIV and adherence-based text messages
  Arms: Multilevel Gaming Adherence
Behavioral: Treatment as Usual + — Combination of electronic medication monitoring device and non-HIV related mobile gaming application
  Arms: Treatment as Usual +

SUMMARY:
Despite the need for consistent adherence to medical care, youth living with HIV have low rates of adherence to medications and treatment. There are few interventions to improve adherence to HIV medications and treatment for youth, and there is a great need for novel approaches that are engaging for this age group. The investigators developed an intervention that includes a mobile gaming app that is integrated with a 7-day electronic medication device and text messages. During gameplay, youth fight HIV in colorful organ systems. A small previous project found that the intervention helped youth who were newly starting medications for HIV by improving adherence and decreasing HIV virus in their bodies (viral load). This proposed project will test the intervention with larger number of youth (100) who are newly starting HIV treatment and medications in New England, Georgia, and in Mississippi. The investigators want to determine if adherence is improved and viral load is reduced in this larger sample.

DETAILED DESCRIPTION:
Despite need for consistent adherence to medical care, youth living with HIV (YLWH) have low rates of adherence and retention in care, and are at great risk for being lost to follow-up.(5,16-18) There is a great need for adherence interventions that are novel and appealing for YLWH.(7,8,14) The investigators developed, and preliminarily examined, a multi-level technology that integrates a 7-day smart medication device WITH an immersive and appealing smartphone app/game that is attractive and engaging for YLWH.(82,83) During gameplay, YLWH fight HIV in colorful and immersive organ systems, and receive adherence related text messages with game graphics. Electronic medication monitoring device openings guide game-related text messages. The investigators tested the Multilevel Gaming Intervention in a developmental trial. The impact of the intervention was greatest among those who had newly begun ART. In participants who had newly begun ART, the intervention decreased viral load and improved ART adherence. Those newly starting ART in the intervention, compared to those newly starting ART in the control, experienced a 0.96 log viral load greater decrease and evidenced a large effect size for improved adherence as measured by an electronic medication monitoring device (d=1.18, 71% vs. 48% adherence at post-test). These interactions between intervention and newly starting ART were significant in ANCOVAs, accounting for baseline values (viral load: F=4.33, p=0.04, adherence: F=3.20, p=0.05). For this next proposed stage of research, the investigators will further test the Multilevel Gaming Intervention with YLWH who are newly starting ART at clinical sites in New England, Georgia, and in Mississippi. A multisite randomized controlled study (48 weeks) among 100 YLWH newly starting ART will test the efficacy of the intervention compared to a control condition (who receive a non-HIV game and the electronic medication monitoring device) on behavioral and biological measures.

ELIGIBILITY:
Inclusion Criteria:

* Living with HIV
* English speaking
* Have started antiretroviral therapy (ART) in the last three months or restarted ART in the last three months after not taking ART for approximately six months
* Have access to a smartphone for the duration of the study
* Not involved with another HIV prevention or adherence related study
* Able to give consent/assent and not impaired by cognitive or medical limitations as per clinical assessment
* Detectable viral load

Exclusion Criteria:

* None

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 107 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Change from Baseline HIV-1 Viral Load at 48 weeks | 48 weeks
  Assessing change from Baseline HIV-1 viral load (copies/mL)

SECONDARY OUTCOMES:
Self-reported Medication Adherence | Baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks
  Proportion of doses taken correctly via electronic pill monitoring device. The proportion of days with correct openings each month will be calculated: (correct openings) / (total number of days in month)
  Assessed at baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks
Self-reported Missed ARV Doses (1 Month) | Baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks
  Proportion of days with missed doses via self-report: (reported missed doses in past month) / (total number of days in month)
  Assessed at baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks
Self-reported Missed ARV Doses (1 week) | Baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks
  Proportion of days with missed doses via self-report: (reported missed doses in past 7 days) / 7
  Assessed at baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks

OTHER OUTCOMES:
HIV Treatment Knowledge Scale | Baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks
  Balfour L, Kowal J, Tasca GA, et al. Development and psychometric validation of the HIV Treatment Knowledge Scale. AIDS Care. 2007;19(9):1141-1148.
  The HIV Treatment Knowledge scale is a 21-item scale that assesses knowledge about complex HIV treatment issues such as co-occurring illnesses and drug resistance. Response options include "True", "False", and "Do not know". Cronbach's alpha was 0.90 in a population of HIV-infected adults. Higher scores indicate greater HIV treatment knowledge.
  Assessed at baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks
Antiretroviral Therapy Treatment Knowledge | Baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks
  The LifeWindows Project Team. The LifeWindows Information Motivation Behavioral Skills ART Adherence Questionnaire (LW-IMB-AAQ). 2006. Center for Health, Intervention, and Prevention. University of Connecticut.
  Antiretroviral therapy treatment knowledge will be assessed with the "Information" subscale from the LifeWindows Information-Motivation-Behavioral Skills ART Adherence Questionnaire. The Information subscale includes 19 Likert-style items. Response options include "Strongly Disagree", "Somewhat Agree", "Neither Agree nor Disagree", "Somewhat Agree", and "Strongly Agree". Cronbach's alpha was 0.60 in a sample of youth living with HIV. Higher scores indicate greater knowledge of ART treatment.
  Assessed at baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks
Motivation for Adherence | Baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks
  The LifeWindows Project Team. The LifeWindows Information Motivation Behavioral Skills ART Adherence Questionnaire (LW-IMB-AAQ). 2006. Center for Health, Intervention, and Prevention. University of Connecticut.
  Motivation for adherence will be assessed with the "Motivation" subscale from the LifeWindows Information-Motivation-Behavioral Skills ART Adherence Questionnaire. The "Motivation" subscale includes 10 Likert-style items that assess personal and social motivations for ART adherence. Cronbach's alpha was 0.75 in a sample of youth living with HIV. Higher scores indicate greater motivation towards adherence.
  Assessed at baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks
Information-Motivation-Behavioral Skills ART Adherence Questionnaire - Behavioral Skills subscale | Baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks
  The LifeWindows Project Team. The LifeWindows Information Motivation Behavioral Skills ART Adherence Questionnaire (LW-IMB-AAQ). 2006. Center for Health, Intervention, and Prevention. University of Connecticut.
  The "Behavioral Skills" subscale from the LifeWindows Information-Motivation-Behavioral Skills ART Adherence Questionnaire assesses perceived ability to perform necessary ART skills. This subscale includes 14 Likert-style items. Response options range from "Very Hard" to "Very Easy". Cronbach's alpha was 0.90 in a sample of youth living with HIV. Higher scores indicate greater motivation towards adherence.
  Assessed at baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks
Medication Adherence Barriers | Baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks
  Simoni JM, Kurth AE, Pearson CR, Pantalone DW, Merrill JO, Frick PA. Self-report measures of antiretroviral therapy adherence: a review with recommendations for HIV research and clinical management. AIDS Behav. 2006; 10(3):227-245. doi: 10.1007/s10461-006-9078-6. PMID: 16783535. PMCID: PMC4083461.
  This 26-item checklist was developed for use by the Adolescent AIDS Trials Network (ATN). This measure assesses common barriers to taking antiretrovirals (ARV) as prescribed and common reasons for stopping ARV.
  Assessed at baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks
Social Support | Baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks
  Martinez J, Harper G, Carleton RA, et al. The Impact of Stigma on Medication Adherence Among HIV-Positive Adolescent and Young Adult Females and the Moderating Effects of Coping and Satisfaction with Health Care. AIDS Patient Care and STDs. 2012;26(2):108-115. doi:10.1089/apc.2011.0178.
  Six Likert-style items assess social support for taking medications, going to medical appointments, and other tasks related to adherence. Responses options range from "Strongly disagree" to "Strongly agree". Cronbach's alpha for this scale is 0.91. Higher scores indicate greater perceived social support.
  Assessed at baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks
HIV Treatment Self-Efficacy | Baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks
  MacDonell KE, Naar-King S, Murphy DA, Parsons JT, Harper GW. Predictors of Medication Adherence in High Risk Youth of Color Living with HIV. Journal of Pediatric Psychology. 2010;35(6):593-601. doi:10.1093/jpepsy/jsp080.
  This six-item, Likert-style scale includes three items that assess self-efficacy for taking medication and three items that assess self-efficacy for adherence to medical appointments. Response options range from "Very Sure I Can" to "Very Sure I Cannot". Higher scores indicate greater self-efficacy for medication and appointment adherence. Cronbach's alpha is 0.92 for this scale.
  Assessed at baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James B Brock, MD, Study Director — University of Mississippi Medical Center; Rachel Epstein, MD, Study Director — Boston Medical Center; Stephen Pelton, MD, Study Director — Boston Medical Center; Larry K Brown, MD, Study Director — Rhode Island Hospital; Laura Whiteley, MD, Principal Investigator — Rhode Island Hospital; Andres Camacho-Gonzalez, MD, Study Director — Emory University
Locations (4):
- United States (4):
  - Emory University, Atlanta, Georgia
  - Boston Medical Center, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Rhode Island Hospital, Providence, Rhode Island

REFERENCES:
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730